CLINICAL TRIAL: NCT02810873
Title: PET Imaging of Breast Cancer Using Oncogene Expression
Brief Title: Positron Emission Tomography Imaging Using Copper Cu 64 TP3805 in Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated by PI
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08F.327; JT 1419 (Other: JeffTrial Number)
Record Dates: First submitted 2016-06-08; First posted 2016-06-23 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Positron-Emission Tomography; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- F-18-FDG Whole body Scan (Experimental): STAGE I: Patients with a positive biopsy and abnormal (positive) fludeoxyglucose F18-labeled PET whole-body scan undergo a whole-body copper Cu 64 TP3805-labeled PET scan.
  Interventions: Device: Positron Emission Mammography; Radiation: Fludeoxyglucose F-18; Drug: Copper Cu 64 TP3805
- No F-18-FDG Scan (Experimental): STAGE II: Patients with a positive biopsy, but no fludeoxyglucose F18 scan undergo a breast fludeoxyglucose F18-labeled PEM Positron Emission Mammography scan followed by a breast copper Cu 64 TP3805-labeled PEM scan.
  Interventions: Device: Positron Emission Tomography; Radiation: Fludeoxyglucose F-18; Drug: Copper Cu 64 TP3805

INTERVENTIONS:
Device: Positron Emission Mammography — Undergo PEM Positron Emission Mammography scan
  Arms: F-18-FDG Whole body Scan
Device: Positron Emission Tomography — Undergo PET Positron Emission Tomography scan
  Other Names: Medical Imaging, Positron Emission Tomography; proton magnetic resonance spectroscopic imaging
  Arms: No F-18-FDG Scan
Radiation: Fludeoxyglucose F-18 — Undergo Fludeoxyglucose F-18 PET (Positron Emission Tomography) /PEM (Positron Emission Mammography) scan
  Other Names: 2-Deoxy-2-(18F)Fluoro-D-Glucose; 2-F18-Fluoro-2-deoxy-D-glucose; 2-F18-Fluoro-2-deoxyglucose; 105851-17-0; 18FDG; 723398; FDG; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Copper Cu 64 TP3805 — Undergo copper Cu 64 TP3805 PET (Positron Emission Tomography) /PEM (Positron Emission Mammography) scan
  Other Names: Cu-64-TP3805

SUMMARY:
This clinical trial studies positron emission tomography imaging in using copper Cu 64 TP3805in patients with breast cancer. Diagnostic procedures, such as positron emission tomography (PET) and positron emission mammography (PEM) scan, using Cu-64-TP3805 may help doctors find and diagnose breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. The study's primary goal is to assess the ability of Cu-64-TP3805 (copper Cu 64 TP3805) to detect primary breast lesions as determined by the F-18-FDG (fludeoxyglucose F 18) scan.

II. The study's second goal is to determine the ability of Cu-64-TP3805 to detect primary breast lesions as determined by histology (sensitivity).

III. The study's third goal is to determine the ability of Cu-64-TP3805 to detect metastatic lesions as identified by the F-18-FDG whole-body scan.

OUTLINE: This is a dose-finding 2-stage study.

STAGE I: Patients with a positive biopsy and abnormal (positive) fludeoxyglucose F18-labeled PET whole-body scan undergo a whole-body copper Cu 64 TP3805-labeled PET scan.

STAGE II: Patients with a positive biopsy, but no fludeoxyglucose F18 scan undergo a breast fludeoxyglucose F18-labeled PEM scan followed by a breast copper Cu 64 TP3805-labeled PEM scan.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Breast cancer shown with abnormal mammogram and histology verification (stage-1 patients will also need to have a positive F-18-FDG whole-body scan)
* Tumor mass of 1 cm or larger, as determined by mammography, ultrasound, or magnetic resonance imaging (MRI)
* Signed informed consent form approved by the institutional review board (IRB)

Exclusion Criteria:

* Pregnant or lactating female
* Patient with asthma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Thakur, PhD, Principal Investigator — Thomas Jefferson University

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- F-18-FDG Whole-body Scan: STAGE I: Patients with a positive biopsy and abnormal (positive) fludeoxyglucose F18-labeled PET whole-body scan undergo a whole-body copper Cu 64 TP3805-labeled PET scan.
- No F-18-FDG Scan: STAGE II: Patients with a positive biopsy, but no fludeoxyglucose F18 scan undergo a breast fludeoxyglucose F18-labeled PEM Positron Emission Mammography scan followed by a breast copper Cu 64 TP3805-labeled PEM scan.
  Positron Emission Mammography: Undergo PEM Positron Emission Mammography scan
  Positron Emission Tomography: Undergo PET Positron Emission Tomography scan
  Fludeoxyglucose F-18: Undergo Fludeoxyglucose F-18 PET (Positron Emission Tomography) /PEM (Positron Emission Mammography) scan
  Copper Cu 64 TP3805: Undergo copper Cu 64 TP3805 PET (Positron Emission Tomography) /PEM (Positron Emission Mammography) scan
Period: Overall Study
Arm/Group | F-18-FDG Whole-body Scan | No F-18-FDG Scan
Started | 6 | 13
Completed | 6 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- F-18-FDG Whole-body Scan: STAGE I: Patients with a positive biopsy and abnormal (positive) fludeoxyglucose F18-labeled PET whole-body scan undergo a whole-body copper Cu 64 TP3805-labeled PET scan.
  Positron Emission Mammography: Undergo PEM Positron Emission Mammography scan
  Positron Emission Tomography: Undergo PET Positron Emission Tomography scan
  Fludeoxyglucose F-18: Undergo Fludeoxyglucose F-18 PET (Positron Emission Tomography) /PEM (Positron Emission Mammography) scan
  Copper Cu 64 TP3805: Undergo copper Cu 64 TP3805 PET (Positron Emission Tomography) /PEM (Positron Emission Mammography) scan
- Total: Total of all reporting groups
Arm/Group | F-18-FDG Whole-body Scan | No F-18-FDG Scan | Total
Number analyzed (Participants) | 6 | 13 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 10 | 16
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 12 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 13 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of F-18-FDG Positive Lesions That Are Detected by the Copper Cu 64 TP3805 Analog
Description: Cu-64 results will be compared with those of F-18-FDG for: The unit of analysis will be the lesion (with potentially multiple lesions available per patient).
Time Frame: 4 hours after Cu 64 TP3805 administered
Measure: Number; unit: Number of Lesions
Arm/Group | F-18-FDG Whole-body Scan | No F-18-FDG Scan
Number analyzed (Participants) | 6 | 13
Number of Lesions | 10 | 14

2. Secondary Outcome: Ability of Copper Cu 64 TP3805 to Detect Primary Breast Lesions as Determined by Histology (Sensitivity)
Description: Optimal imaging time is the one (of the three) which will have least background activity in the surrounding tissue and image the maximum number of lesions with clarity. 95% confidence intervals will be used. To account for the multiplicity of lesions per patient, the GEE approach will be used, with the robust variance. Any adverse events will be summarized descriptively.
Time Frame: 4 hours after Cu 64 TP3805 administered
Population: No data were collected or reported as tumors were not extracted and histology could not be performed
Arm/Group | F-18-FDG Whole-body Scan | No F-18-FDG Scan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | F-18-FDG Whole-body Scan | No F-18-FDG Scan
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/13
Other Adverse Events (participants affected / at risk) | 0/6 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-18-FDG Whole-body Scan (N=6) | No F-18-FDG Scan (N=13)
Flushing sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes